CLINICAL TRIAL: NCT02232165
Title: Mean Arterial Pressure in Spinal Cord Injury (MAPS): Determination of Non-inferiority of a Mean Arterial Pressure Goal of 65 mmHg Compared to a Mean Arterial Pressure Goal of 85 mmHg in Acute Human Traumatic Spinal Cord Injury.
Brief Title: Mean Arterial Blood Pressure Treatment for Acute Spinal Cord Injury
Acronym: MAPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Hotchkiss Brain Institute, University of Calgary (Other); AANS/CNS Section on Disorders of the Spine and Peripheral Nerves (Other)
Responsible Party: Principal Investigator, Dr W. Bradley Jacobs, Assistant Professor, Department of Clinical Neurosciences, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-24927
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Acute Spinal Cord Injury
Keywords: acute spinal cord injury; hemodynamic therapy; functional outcome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypotension avoidance (MAP >= 65 mmHg) (Experimental): Mean arterial blood pressure is maintained >= 65 mmHg for 7 days following acute SCI.
  Interventions: Other: Hypotension avoidance
- Induced hypertension (MAP >= 85 mmHg) (Active Comparator): Induced hypertension with mean arterial blood pressure >= 85 mmHg for 7 days following acute SCI.
  Interventions: Other: Induced hypertension

INTERVENTIONS:
Other: Hypotension avoidance — Induced hypertension with MAP >= 85 mmHg for 7 days following SCI is the current recommended clinical option guideline. Our intervention tests whether hypotension avoidance and maintenance of MAP >= 65 mmHg is not inferior to induced hypertension.
  Arms: Hypotension avoidance (MAP >= 65 mmHg)
Other: Induced hypertension — Induced hypertension with MAP >= 85 mmHg for 7 days following SCI is the current recommended clinical option guideline.
  Arms: Induced hypertension (MAP >= 85 mmHg)

SUMMARY:
Current guidelines for the clinical management of acute spinal cord injury (SCI) recommend maintenance of mean arterial blood pressure (MAP) at 85 to 90 mmHg for the first seven days after SCI as a clinical option. Unfortunately, the medical evidence to support this recommendation exists only at the clinical case series level (Class III data). Furthermore, maintenance of sustained systemic hypertension, as per clinical guidelines, may be associated with risks to the patient via adverse medical events. Given this equivocal evidence, the investigators group has questioned the merit of sustained induced hypertension following acute SCI and has previously conducted a randomized, prospective controlled feasibility study to further examine this issue. This prior pilot study randomized patients with acute SCI to a spinal cord perfusion pressure (SCPP = MAP - intrathecal pressure (ITP)) target of ≥ 75 mmHg or to a control group (hypotension avoidance, MAP ≥ 65 mmHg). The primary endpoint measure was defined as the change in American Spinal Injury Association (ASIA) motor score from baseline. No difference in the primary outcome was noted at one-year post-SCI in this study.

In light of this pilot data, the investigators hypothesize that maintenance of normotension (MAP ≥ 65mmHg) is not inferior to induced hypertension (MAP ≥ 85mmHg) for 7 days following acute SCI. As such, the investigators propose to conduct a Phase III non-inferiority prospective, randomized clinical trial in acute SCI patients. Subjects will be randomized into one of two MAP management groups for 7 days; Group 1 will be managed with a target MAP ≥ 65 mmHg, while Group 2 will be managed with a target MAP ≥ 85 mmHg. The primary endpoint will be change in ASIA motor score from baseline at 12 months post injury. A difference of ≤10 ASIA motor points change from baseline between groups will be considered as non-inferiority. Secondary endpoints will include ASIA sensory score, proportion of patients achieving a one grade improvement in ASIA impairment scale, quality of life assessment (as measured by Short-Form-36 [SF-36]) and functional outcome (as measured by the Spinal Cord Independence Measure (SCIM) and Functional Independence Measure (FIM). These will be measured at baseline, 72 hours and 3, 6 and 12 months from injury. Adverse events will be meticulously recorded. The information gleaned from this trial will provide valuable information for the acute treatment of traumatic SCI and will serve the objective of optimizing current clinical practice and thus maximizing medical and neurological outcome for individuals following acute traumatic SCI.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 16 years.
* Motor complete or incomplete (ASIA A, B, or C) acute traumatic SCI involving spinal levels between C0 and T12.
* Written and informed consent from patient or a legally acceptable representative.
* Randomization and initiation of management protocol within 24 hours of injury.
* Reasonable expectation of availability to receive the full 7-day course of therapy and be available for follow up evaluations.

Exclusion Criteria:

* Acute traumatic SCI > 24 hours old.
* Central cord syndrome, defined as ASIA C or D with mean lower extremity score greater than upper extremity score.
* Isolated sensory deficit, motor intact.
* Isolated radicular motor deficit, defined as a unilateral motor deficit restricted to a single myotome.
* Pregnancy.
* Associated conditions interfering with informed consent or outcome assessment including closed head injury and major orthopedic injuries.
* Polytrauma: Abbreviated Injury Severity Score >3 in any area other than head.
* Known uncorrected severe coronary artery disease or evidence of active coronary ischemia (ECG changes, positive troponin) will be excluded.
* Advanced cardiac, pulmonary, hepatic or liver disease; the former will be operationally defined using NCI Toxicity Criteria (Grade 2 or higher).
* Allergy or other contraindication to norepinephrine.
* A known diagnosis of cancer (except basal cell cancer).
* Uncontrolled hypertension, defined as blood pressure persistently above 220 mmHg systolic or 120 mmHg diastolic, despite antihypertensive therapy.
* Any patients living in a nursing home or supervised living centre. Patients must be historically fully independent in all activities of daily living including banking, shopping, cooking, toileting, showering and dressing.
* Any other medical condition, in the investigator's opinion, for which the patient should not be included in the trial.
* Pre-existing and active major psychiatric or other chronic neurological disease.
* Patients who have a history of substance abuse or dependency within 12 months prior to the study.
* Currently participating in another interventional investigational study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-02; Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Change in ASIA motor score from baseline | 1 year post-injury
  A difference of ≤10 ASIA motor points change from baseline between groups will be considered as non-inferiority.

SECONDARY OUTCOMES:
ASIA sensory score | 1 year post-injury
Proportion of patients achieving a one-grade improvement in ASIA impairment scale (AIS) | 1 year post-injury
Quality of life assessment with Short-Form-36 (SF-36) | 1 year post-injury
Functional outcome assessment with FIM and SCIM | 1 year post-injury

OTHER OUTCOMES:
Number and severity of adverse events | Within 1 year of study enrolment

CONTACTS AND LOCATIONS:
Overall Officials: W. Bradley Jacobs, MD, Principal Investigator — University of Calgary
Locations (2):
- University of Texas Health Science Center San Antonio, San Antonio, Texas, United States
- University of Calgary, Foothills Medical Centre, Calgary, Alberta, Canada